CLINICAL TRIAL: NCT03159468
Title: Alcohol-Related Sexual Aggression: An Emotion Regulation Intervention
Brief Title: Emotion Regulation Interventions for Alcohol-Related Sexual Aggression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Arizona State University (Other)
Responsible Party: Principal Investigator, Kelly Cue Davis, Associate Professor, University of Washington
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00002103; 1R21AA023811-01A1 (NIH)
Record Dates: First submitted 2017-05-12; First posted 2017-05-18 (Actual); Results first posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Sexual Aggression; Heavy Drinking
MeSH Terms: interventions — Cognitive Restructuring; Mindfulness; Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cognitive Restructuring & Alcohol Condition (Experimental): Participants will receive a brief online training regarding the use of cognitive restructuring skills to cope with negative emotions. They will then consume an alcoholic beverage in the lab.
  Interventions: Behavioral: Cognitive Restructuring; Other: Alcohol consumption
- Mindfulness & Alcohol Condition (Experimental): Participants will receive a brief online training regarding the use of mindfulness skills to cope with negative emotions. They will then consume an alcoholic beverage in the lab.
  Interventions: Behavioral: Mindfulness; Other: Alcohol consumption
- Nutrition Information & Alcohol Condition (Experimental): Participants will receive general information about nutrition. They will then consume an alcoholic beverage in the lab.
  Interventions: Other: Alcohol consumption
- Cognitive Restructuring & No Alcohol Condition (Experimental): Participants will receive a brief online training regarding the use of cognitive restructuring skills to cope with negative emotions. They will then consume a non-alcoholic beverage in the lab.
  Interventions: Behavioral: Cognitive Restructuring
- Mindfulness & No Alcohol Condition (Experimental): Participants will receive a brief online training regarding the use of mindfulness skills to cope with negative emotions. They will then consume a non-alcoholic beverage in the lab.
  Interventions: Behavioral: Mindfulness
- Nutrition Information & No Alcohol Condition (No Intervention): Participants will receive general information about nutrition. They will then consume a non-alcoholic beverage in the lab.

INTERVENTIONS:
Behavioral: Cognitive Restructuring — Participants receive didactic instruction regarding cognitive restructuring skills and then practice using these skills in hypothetical situations.
  Arms: Cognitive Restructuring & Alcohol Condition; Cognitive Restructuring & No Alcohol Condition
Behavioral: Mindfulness — Participants receive didactic instruction regarding mindfulness skills and then practice using these skills in hypothetical situations.
  Arms: Mindfulness & Alcohol Condition; Mindfulness & No Alcohol Condition
Other: Alcohol consumption — Participants consume an alcoholic beverage in the lab.
  Arms: Cognitive Restructuring & Alcohol Condition; Mindfulness & Alcohol Condition; Nutrition Information & Alcohol Condition

SUMMARY:
Rates of sexual assault are alarmingly high, and alcohol is consistently implicated in the majority of these assaults. Despite well-intentioned prevention efforts, this pandemic continues unabated, warranting the development of novel and innovative approaches to the reduction of sexual aggression. The goal of this research is to evaluate the efficacy of two brief online emotion regulation interventions for reducing alcohol-related sexual aggression in heavy episodic drinking young men with a sexual aggression history. Previous research suggests that emotion regulation difficulties are associated with both alcohol consumption and aggressive behavior. Despite the potential prevention utility of improving sexually aggressive men's emotion regulation skills in order to reduce their alcohol-related sexual aggression, this approach has yet to be explored. Thus, this study evaluates the effects of two brief online ER interventions - cognitive restructuring and mindfulness - on men's emotion regulation during a sexual aggression-related analogue. Additionally, these effects will be evaluated during both sober and intoxicated states through a laboratory- based alcohol administration experiment.

ELIGIBILITY:
Inclusion Criteria:

* Single
* Male
* Age 21-30
* Heterosexually active within past year
* Heavy episodic drinker
* Self-reported history of sexual aggression

Exclusion Criteria:

* History of alcohol problems
* Medical condition or medications that contraindicate alcohol consumption

Ages: 21 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Self-defined as male
Enrollment: 209 (Actual)
Dates: Start 2016-12-31 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-06-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All enrolled participants were assigned to one of the six arms.
Groups:
- Cognitive Restructuring & Alcohol Condition: Participants will receive a brief online training regarding the use of cognitive restructuring skills to cope with negative emotions, then consume an alcoholic beverage in the lab.
  Cognitive Restructuring: Participants receive didactic instruction regarding cognitive restructuring skills and then practice using these skills in hypothetical situations.
- Mindfulness & Alcohol Condition: Participants will receive a brief online training regarding the use of mindfulness skills to cope with negative emotions, then receive an alcoholic beverage in the lab.
  Mindfulness: Participants receive didactic instruction regarding mindfulness skills and then practice using these skills in hypothetical situations.
- Nutrition Information & Alcohol Condition: Participants receive general information about nutrition, then receive an alcoholic beverage in the lab.
- Cognitive Restructuring & No Alcohol Condition: Participants will receive a brief online training regarding the use of cognitive restructuring skills to cope with negative emotions, then consume a non-alcoholic beverage in the lab.
  Cognitive Restructuring: Participants receive didactic instruction regarding cognitive restructuring skills and then practice using these skills in hypothetical situations.
- Mindfulness & No Alcohol Condition: Participants will receive a brief online training regarding the use of mindfulness skills to cope with negative emotions, then receive a non-alcoholic beverage in the lab.
  Mindfulness: Participants receive didactic instruction regarding mindfulness skills and then practice using these skills in hypothetical situations.
- Nutrition Information & No Alcohol Condition: Participants receive general information about nutrition, then receive a non-alcoholic beverage in the lab.
Period: Overall Study
Arm/Group | Cognitive Restructuring & Alcohol Condition | Mindfulness & Alcohol Condition | Nutrition Information & Alcohol Condition | Cognitive Restructuring & No Alcohol Condition | Mindfulness & No Alcohol Condition | Nutrition Information & No Alcohol Condition
Started | 35 | 35 | 37 | 34 | 34 | 34
Completed | 35 | 35 | 34 | 34 | 34 | 34
Not Completed | 0 | 0 | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cognitive Restructuring & Alcohol Condition: Participants received a brief online training regarding the use of cognitive restructuring skills to cope with negative emotions, then received an alcoholic beverage in the lab.
  Cognitive Restructuring: Participants receive didactic instruction regarding cognitive restructuring skills and then practice using these skills in hypothetical situations.
- Mindfulness & Alcohol Condition: Participants received a brief online training regarding the use of mindfulness skills to cope with negative emotions, then received an alcoholic beverage in the lab.
  Mindfulness: Participants receive didactic instruction regarding mindfulness skills and then practice using these skills in hypothetical situations.
- Nutrition Information & Alcohol Condition: Participants received general information about nutrition, then received an alcoholic beverage in the lab.
- Cognitive Restructuring & No Alcohol Condition: Participants received a brief online training regarding the use of cognitive restructuring skills to cope with negative emotions, then received a non-alcoholic beverage in the lab.
  Cognitive Restructuring: Participants receive didactic instruction regarding cognitive restructuring skills and then practice using these skills in hypothetical situations.
- Mindfulness & No Alcohol Condition: Participants received a brief online training regarding the use of mindfulness skills to cope with negative emotions, then received a non-alcoholic beverage in the lab.
  Mindfulness: Participants receive didactic instruction regarding mindfulness skills and then practice using these skills in hypothetical situations.
- Nutrition Information & No Alcohol Condition: Participants received general information about nutrition, then received a non-alcoholic beverage in the lab.
- Total: Total of all reporting groups
Arm/Group | Cognitive Restructuring & Alcohol Condition | Mindfulness & Alcohol Condition | Nutrition Information & Alcohol Condition | Cognitive Restructuring & No Alcohol Condition | Mindfulness & No Alcohol Condition | Nutrition Information & No Alcohol Condition | Total
Number analyzed (Participants) | 35 | 35 | 37 | 34 | 34 | 34 | 209
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.67 (2.88) | 24.06 (2.78) | 25.09 (3.03) | 25.32 (2.58) | 24.35 (2.60) | 25.08 (2.68) | 24.76 (2.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 35 | 35 | 37 | 34 | 34 | 34 | 209
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 3 | 3 | 6 | 3 | 21
  Not Hispanic or Latino | 33 | 31 | 34 | 31 | 28 | 30 | 187
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 5 | 8 | 6 | 7 | 7 | 37
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 4 | 2 | 0 | 2 | 5 | 14
  White | 26 | 22 | 18 | 25 | 18 | 16 | 125
  More than one race | 3 | 4 | 6 | 2 | 4 | 4 | 23
  Unknown or Not Reported | 1 | 0 | 3 | 1 | 3 | 2 | 10
Body Weight [Mean (Standard Deviation); unit: pounds] | 175.29 (26.54) | 170.34 (24.66) | 170.26 (26.75) | 184.09 (48.79) | 173.53 (21.29) | 170.97 (21.00) | 174.07 (29.72)

OUTCOME MEASURES:

1. Primary Outcome: Sexual Aggression Intentions
Description: Sexual Aggression Intentions Scale. Construct: Self-reported ratings of sexual aggression likelihood in a hypothetical scenario. Minimum value of 1 ("Very unlikely"). Maximum value of 7 ("Very likely"). Higher scores mean a worse outcome.
Time Frame: Within one hour after receiving the intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Restructuring & Alcohol Condition | Mindfulness & Alcohol Condition | Nutrition Information & Alcohol Condition | Cognitive Restructuring & No Alcohol Condition | Mindfulness & No Alcohol Condition | Nutrition Information & No Alcohol Condition
Number analyzed (Participants) | 35 | 35 | 34 | 34 | 34 | 34
score on a scale | 1.58 (1.12) | 1.90 (1.28) | 2.18 (1.59) | 1.53 (1.16) | 1.38 (.90) | 1.70 (1.15)
Statistical Analysis 1: Comparison: Cognitive Restructuring & Alcohol Condition vs Mindfulness & Alcohol Condition vs Nutrition Information & Alcohol Condition vs Cognitive Restructuring & No Alcohol Condition vs Mindfulness & No Alcohol Condition vs Nutrition Information & No Alcohol Condition; Test type: Other; p = .041, ANOVA — This p-value is for the main effect of beverage condition
Statistical Analysis 2: Comparison: Cognitive Restructuring & Alcohol Condition vs Mindfulness & Alcohol Condition vs Nutrition Information & Alcohol Condition vs Cognitive Restructuring & No Alcohol Condition vs Mindfulness & No Alcohol Condition vs Nutrition Information & No Alcohol Condition; Test type: Other; p = .160, ANOVA — This p-value is for the main effect of intervention condition
Statistical Analysis 3: Comparison: Cognitive Restructuring & Alcohol Condition vs Mindfulness & Alcohol Condition vs Nutrition Information & Alcohol Condition vs Cognitive Restructuring & No Alcohol Condition vs Mindfulness & No Alcohol Condition vs Nutrition Information & No Alcohol Condition; Test type: Other; p = .462, ANOVA — This p-value is for the beverage condition by intervention condition interaction

ADVERSE EVENTS:
Time Frame: During the in-lab study experiment. There was no follow-up period.
Groups:
- Cognitive Restructuring & Alcohol Condition: Participants will receive a brief online training regarding the use of cognitive restructuring skills to cope with negative emotions, then receive an alcoholic beverage.
  Cognitive Restructuring: Participants receive didactic instruction regarding cognitive restructuring skills and then practice using these skills in hypothetical situations.
- Mindfulness & Alcohol Condition: Participants will receive a brief online training regarding the use of mindfulness skills to cope with negative emotions, then receive an alcoholic beverage.
  Mindfulness: Participants receive didactic instruction regarding mindfulness skills and then practice using these skills in hypothetical situations.
- Nutrition Information & Alcohol Condition: Participants will receive general information about nutrition, then receive an alcoholic beverage.
- Cognitive Restrucuring & No Alcohol Condition: Participants will receive a brief online training regarding the use of cognitive restructuring skills to cope with negative emotions, then receive a non-alcoholic beverage.
  Cognitive Restructuring: Participants receive didactic instruction regarding cognitive restructuring skills and then practice using these skills in hypothetical situations.
- Mindfulness & No Alcohol Condition: Participants will receive a brief online training regarding the use of mindfulness skills to cope with negative emotions, then receive a non-alcoholic beverage.
  Mindfulness: Participants receive didactic instruction regarding mindfulness skills and then practice using these skills in hypothetical situations.
- Nutrition Information & No Alcohol Condition: Participants will receive general information about nutrition, then receive a non-alcoholic beverage.
Arm/Group | Cognitive Restructuring & Alcohol Condition | Mindfulness & Alcohol Condition | Nutrition Information & Alcohol Condition | Cognitive Restrucuring & No Alcohol Condition | Mindfulness & No Alcohol Condition | Nutrition Information & No Alcohol Condition
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35 | 0/37 | 0/34 | 0/34 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35 | 0/37 | 0/34 | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35 | 0/37 | 0/34 | 0/34 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-16): https://cdn.clinicaltrials.gov/large-docs/68/NCT03159468/Prot_SAP_000.pdf